CLINICAL TRIAL: NCT06352008
Title: To Evaluate the Efficacy and Safety of Anlotinib Hydrochloride Capsule in Postoperative Non-pCR Patients With Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20230553
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experiment (Experimental)
  Interventions: Drug: Anlotinib

INTERVENTIONS:
Drug: Anlotinib — 12mg once a day, taken orally before breakfast for 2 consecutive weeks and stopped for 1 week. Without special circumstances, it is recommended to take at a fixed time every day; If there is a missing dose during the administration, confirm that the time before the next administration is less than 12 hours, no more refilling. The maximum duration of drug use is tentatively 1 year.

SUMMARY:
To explore the effectiveness of anlotinib hydrochloride capsule in postoperative non-pCR non-small cell lung cancer patients with adjuvant intensive therapy

ELIGIBILITY:
Inclusion Criteria:

1. The subjects voluntarily joined the study, signed the informed consent, and the compliance was good;
2. ≥18 years old (calculated by the date of signing the informed consent); Both men and women; ECOG score 0~1; Expected survival ≥3 months;
3. Patients with stage IIA-IIIA NSCLC who had previously received PD-1/PD-L1 inhibitors combined with chemotherapy neoadjuvant therapy and underwent R0 resection for curative purposes before surgery (note: the disease was presented in the American Joint Committee on Cancer (AJCC)/Union International Against Cancer (UICC) 8th edition of lung cancer TNM staging);
4. For patients who did not achieve pathological complete response after PD-1/PD-L1 inhibitor combined with chemotherapy neoadjuvant treatment, and the time between the first trial medication after surgery was required to be 4-12 weeks;
5. The main organs function well and meet the standards;
6. Women of reproductive age should agree that effective contraception must be used during the study period and for 6 months after the end of the study, and that serum or urine pregnancy tests are negative within 7 days prior to study enrollment; Men should agree that effective birth control must be used during the study period and for 6 months after the end of the study period.

Exclusion Criteria:

1. Have had or are currently suffering from other malignant tumors within 5 years. The following two conditions can be included: other malignancies treated with a single operation, achieving continuous 5-year disease-free survival (DFS); Cured cervical carcinoma in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (non-invasive tumor), Tis (cancer in situ) and T1 (tumor infiltrating basal membrane)];
2. Subjects are known to have genetic abnormalities that have been approved for targeted drug therapy (non-squamous cell carcinoma subjects are required to have EGFR or ALK gene tested or provide previous test reports during the screening period)
3. Cardiovascular and cerebrovascular abnormalities:

   1. Patients with past or existing heart failure, degree II or higher heart block;
   2. Past or present myocardial infarction or unstable angina pectoris, clinically significant supraventricular or ventricular arrhythmias requiring treatment or intervention;
   3. Occurrence of arteriovenous thrombosis/cancer embolus events within 6 months, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction requiring clear diagnosis), vascular embolism (including deep vein thrombosis, arterial thrombosis, pulmonary embolism, etc.);
4. Participated in other drug clinical trials within the past 30 days;
5. Within 2 weeks before starting the administration, it has been treated with Chinese patent medicines (including compound Cantharides capsule, Kangai injection, Kanglaite capsule/injection, Aidi injection, Bruceae oil injection/capsule, Xiaoaipingtablet/injection, hualbufatin capsule, etc.) with anti-tumor indications specified in the NMPA approved drug instructions;
6. Received major surgery other than radical resection of lung cancer within 4 weeks prior to initiation of administration; According to the investigator, the patient was not eligible to participate in this clinical study for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Event-Free Survival (EFS) | 2 years
  Defined as the time from the first dose administration to the occurrence of any of the following "events": 1. Non-small cell lung cancer recurrence/metastasis confirmed by pathology or imaging; 2. Disease progression; 3. All-cause death (whichever occurs first).

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute & Hospital, Tianjin, China